CLINICAL TRIAL: NCT03906578
Title: Effect of a Probiotic on Blood Pressure in Low-to-moderate Risk Grade 1 Hypertension - a Randomized Study
Brief Title: Effects of a Probiotic in Hypertension
Acronym: HYPRO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Kristin Kraeker, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HYPRO
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Two sachets Vivomixx® containing 8 strains of life bacteria (9 x 10^11 CFU) in the evening for 8 weeks
  Interventions: Dietary Supplement: Vivomixx®
- Placebo (Placebo Comparator): Two sachets placebo in the evening for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vivomixx® — Microbiotic food supplement with L. paracasei, L. plantarum, L. acidophilus, L. delbrueckii, B. longum, B. infantis, B. breve, S. thermophilus
  Arms: Probiotic
Other: Placebo — Placebo with similar appearance to probiotic
  Arms: Placebo

SUMMARY:
High blood pressure is a major risk factor for cardiovascular events, including stroke, heart and kidney failure. Typical anti-hypertensive drugs target vessels, the kidneys or the heart. Here we propose a randomized, placebo-controlled study to test the blood pressure-lowering effect of a probiotic in 110 patients with grade 1 hypertension. In addition, we will investigate glucose variability, fecal bacterial metabolome, peripheral blood effector T cell frequencies (%) and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women
* Treated or untreated hypertension (resting office blood pressure 130-159/80-99 mmHg)
* BMI 18.5 - 34.9 kg/m^2

Exclusion Criteria:

* Secondary causes of hypertension
* Known target organ damage
* 10 years cardiovascular risk score of >20%
* Diabetes
* Established cardiovascular or renal disease
* Other serious diseases
* Recent use of antibiotics
* Specialized diets, e.g. use of probiotics

Comments:

* Two inclusion criteria were changed in June 2021 to improve recruitment
* Age was changed from 50-75 to 50-80 years
* Resting blood pressure was changed from 140-159/90-99 to 130-159/80-99 mmHg

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Nocturnal systolic blood pressure | After 8 weeks compared to placebo and adjusted to baseline
  Measured by 24h ABPM (mmHg)

SECONDARY OUTCOMES:
Nocturnal diastolic blood pressure | After 8 weeks compared to placebo and adjusted to baseline
  Measured by 24h ABPM (mmHg)
24h systolic blood pressure | After 8 weeks compared to placebo and adjusted to baseline
  Measured by 24h ABPM (mmHg)
24h diastolic blood pressure | After 8 weeks compared to placebo and adjusted to baseline
  Measured by 24h ABPM (mmHg)
Office systolic blood pressure | After 8 weeks compared to placebo and adjusted to baseline
  Mean of five consecutive blood pressure measurements (mmHg)
Office diastolic blood pressure | After 8 weeks compared to placebo and adjusted to baseline
  Mean of five consecutive blood pressure measurements (mmHg)
Reduction of antihypertensive medication | After 8 weeks compared to placebo and adjusted to baseline
  Number and dosage of prescribed medication
Glucose variability after standardized breakfasts | After 8 weeks compared to placebo and adjusted to baseline
  Measured by continuous glucose monitoring
Gut microbiome | After 8 weeks compared to placebo and adjusted to baseline
  Change of fecal microbiome composition
Metabolomics stool and serum | After 8 weeks compared to placebo and adjusted to baseline
  Change of fecal and serum metabolome
Change in immune cell phenotypes | After 8 weeks compared to placebo and adjusted to baseline
  Peripheral blood effector T cell frequencies (%)
PROMIS-29 domain pain interference | After 8 weeks compared to placebo and adjusted to baseline
  Range 0-10 with 0 indicating no pain
PROMIS-29 domain depression | After 8 weeks compared to placebo and adjusted to baseline
  Lower (better) T-score (mean 50, SD 10)
PROMIS-29 domain anxiety | After 8 weeks compared to placebo and adjusted to baseline
  Lower (better) T-score (mean 50, SD 10)
PROMIS-29 domain physical function | After 8 weeks compared to placebo and adjusted to baseline
  Higher (better) T-score (mean 50, SD 10)
PROMIS-29 domain fatigue | After 8 weeks compared to placebo and adjusted to baseline
  Lower (better) T-score (mean 50, SD 10)
PROMIS-29 domain sleep disturbance | After 8 weeks compared to placebo and adjusted to baseline
  Lower (better) T-score (mean 50, SD 10)
PROMIS-29 domain ability to participate in social roles and activities | After 8 weeks compared to placebo and adjusted to baseline
  Higher (better) T-score (mean 50, SD 10)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Mähler, PhD, Principal Investigator — Charite University, Berlin, Germany; Dominik N. Müller, PhD, Principal Investigator — Max Delbruck Center (MDC); Ralf Dechend, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Experimental and Clinical Research Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of reported articles (text, tables, figures, supplemental data) will be shared after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Mahler A, Wilck N, Rauch G, Dechend R, Muller DN. Effect of a probiotic on blood pressure in grade 1 hypertension (HYPRO): protocol of a randomized controlled study. Trials. 2020 Dec 29;21(1):1032. doi: 10.1186/s13063-020-04973-0. PMID 33375942
- See also: Protocol publication — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-020-04973-0